CLINICAL TRIAL: NCT03312153
Title: Effect of Neem (Azadirachta Indica) Versus 2.5% Sodium Hypochlorite as Root Canal Irrigants on the Intensity of Post-operative Pain and Amount of Endotoxins in Necrotic Teeth
Brief Title: Effect of Neem and NaOCl on Postoperative Pain and Amount of Endotoxins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadia Saeed Hosny, Nadia Hosny, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Irrigants in endodontics
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Pain; Postoperative Pain; Postoperative Complications; Necrosis; Pathologic Processes
MeSH Terms: conditions — Pain; Pain, Postoperative; Postoperative Complications; Necrosis; Pathologic Processes | interventions — neem oil; Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: * The study will be double-blinded which are the patients and the assessor.
  * The participants will drag the envelop and will not know which irrigant they will be treated with to not affect their behavior and their responses to the subjective outcome measures. also, not provide biased assessment of the effectiveness of the intervention .
  * The study will be double-blinded which are the patients and the assessor.
  * The participants will drag the envelop and will not know which irrigant they will be treated with .
  * Assessors in the microbiology laboratory in Microbiology department, Faculty of Medicine, Cairo University also will be blinded during assessment of data of endotoxins will not know the treatment group of the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neem (Azadirachta indica) (Experimental): Neem (Azadirachta indica) (alcoholic solution) used as an anti inflammatory , antibacterial irrigant
  Interventions: Drug: Neem
- 2.5%sodium hypochlorite (Active Comparator): 2.5% sodium hypochlorite, anti-bacterial root canal irrigant solution
  Interventions: Drug: 2.5% sodium hypochlorite

INTERVENTIONS:
Drug: Neem — A natural irrigant solution act as anti-inflammatory and anti bacterial
  Other Names: Azadirachta indica
  Arms: Neem (Azadirachta indica)
Drug: 2.5% sodium hypochlorite — anti bacterial root canal irrigant solution
  Other Names: 2.5% NaOCL
  Arms: 2.5%sodium hypochlorite

SUMMARY:
The aim of this study is to compare the effect of Neem (azadirachta indica) and 2.5% sodium hypochlorite as root canal irrigants on the intensity of post-operative pain and the amount of endotoxins in necrotic teeth.

DETAILED DESCRIPTION:
According to the eligibility and exclusion criteria the patients will be selected and randomly divided into two groups. The operator N.S. will complete endodontic treatment of all cases in two visits as following:

1. Anaesthetizing the tooth using inferior alveolar nerve block followed by buccal infiltration technique.
2. Isolation the tooth with a rubber dam and disinfect the tooth using sterile swabs moistened with 30% H2O2 (v/v) for 30 seconds followed by 5.25% NaOCl for 30 seconds and 5% sodium thiosulphate for inactivation of the disinfecting agents .
3. Performing access cavity preparation in two stage :

   1. The first stage: will be performed to allow removal of contamination which includes carious lesions and restoration using high speed sterile round bur and diamond stone.
   2. In second stage: before entering the pulp chamber, the access cavity will be disinfected .
4. For endotoxins sampling, the first sample (S1):

   N.S. will take the sample by introducing a sterile paper point (size #15) into the full working length of the wider / largest canals or canals that show presence of the exudate.
5. N.S. will place the sample in a sterile glass for further Enzyme-linked immunosorbent assay (ELISA).
6. After the first sampling,Taking working length using electronic apex locator and then will be confirmed radio-graphically .
7. Performing the biomechanical preparation for the two groups in a crown-down technique using ProTaper Next rotary system.
8. Irrigation with 2mL of specified irrigation either 2.5% NaOCl or Neem irrigant will be performed each time instrument is changed with 30-gauge side-vented needles.
9. After complete mechanical preparation, the root canals will be flushed using 5mL of sterile saline solution.
10. Before the second sampling (S2):

    N.S. will irrigate the prepared root canal with 5 mL of 17% EDTA solution for 3 minutes followed by a final rinse with 5 mL of a sterile saline solution to remove smear layer. NS will seal the access cavity with temporary filling material.
11. Scheduling the second appointment 1 week after the first appointment;. NS will irrigate the root canals with 5 mL of a sterile saline solution.
12. N.S. will give the patients a pain diary to record the postoperative pain after 6,12,24 and 48h post-instrumentation.
13. in second appointment: After master cone fit radiograph and selection of the master cone, all canals will be filled using cold lateral condensation technique with resin-based sealer.
14. N.S. will give the patients another pain diary to record the postoperative pain after 6, 12, 24 and 48 hours post-obturation.

ELIGIBILITY:
Inclusion Criteria:

* 1- Mandibular molar teeth:

  * Diagnosed clinically with pulp necrosis.
  * Absence of spontaneous pain
  * Pain on palpation or tenderness to percussion.
  * Periradicular radiolucency or widening of periodontal membrane space. 2- Patients' acceptance to participate in the trial. 3- Patients who can understand NRS scale and can sign the informed consent.

Exclusion Criteria:

* 1. Primary teeth and permanent teeth with immature roots which require special endodontic treatment protocol that seeking for obtaining good apical seal, proper cleaning, shaping and obturation 2. Patients who have received antibiotics for the last 3 months before the study or any medication that could alter their perception of pain, inflammation and infection .

  3. Teeth previously accessed or endodontically treated as they have low success rate .

  4. Patients with diabetes, immune-compromising and immune-suppresion disease as the healing is much more slowly and more liable to infection .

  5. Pregnant patients to avoid exposure to radiograph. Moreover, pain perception may be altered due to hormonal changes .

  6. Teeth with deep pocket >4 mm as it has poor prognosis and deep pockets are harbor area for infection which need specific surgical and periodontal treatment .

  7. Teeth that could not be isolated with a rubber-dam or could not be restorable.

  8. Tooth associated with vertical root fracture, coronal perforation, calcification and external or internal root resorption as it has poor prognosis.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
post operative pain | Up to 48 hours
  post-instrumentaion pain and post-instrumentation pain assessed with the Numerical Rating Pain Scale

SECONDARY OUTCOMES:
endotoxins | 6 hours
  The quantitative enzyme-linked immunosorbent assay (ELISA) is a plate-based assay technique and is considered highly sensitive and specific test for detection and quantifying of endotoxin in the root canals by using a commercial standard kit. The samples will be collected by the operator and will be stored at -80C so that all the samples would be processed at the same time by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided